CLINICAL TRIAL: NCT04720482
Title: The Capacity of Neurological Pupil Index to Predict the Absence of Somatosensory Evoked Potentials in Comatose Survivors of Cardiac Arrest
Brief Title: Pupillometry and Somatosensory Evoked Potential in Cardiac Arrest
Acronym: PASCA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Christian Rylander, Associate Professor, Sahlgrenska University Hospital
Other Study IDs: PASCA
Record Dates: First submitted 2020-09-05; First posted 2021-01-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Arrest; Cardiopulmonary Arrest With Successful Resuscitation; Resuscitation
MeSH Terms: conditions — Heart Arrest | interventions — Evoked Potentials, Somatosensory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Comatose survivors of cardiac arrest: Adult (>18 years) patients remaining comatose during intensive care 48 hours after cardiac arrest. All patients are submitted to both clinical routine measurements: pupillometry and somatosensory evoked potentials.
  Interventions: Diagnostic Test: Somatosensory Evoked Potentials; Diagnostic Test: Automated Pupillometry

INTERVENTIONS:
Diagnostic Test: Somatosensory Evoked Potentials — SSEP performed bilaterally with stimulation of the median nerve
  Other Names: Cortical N20 response
Diagnostic Test: Automated Pupillometry — PLR quantified as NPi using a handheld automated pupillometer
  Other Names: Neurological Pulpil index

SUMMARY:
Somatosensory Evoked Potentials (SSEP) and Pupillary Light Reflex (PLR) are key methods for neurologic prognostication in comatose survivors of cardiac arrest. Both methods have low false positive rates.Though they assess different functions of the brain, they should both be sensitive to severe anoxic/ischemic injury from cardiac arrest. The aim of this observational prospective study with an estimated recruitment of 50 patients is to examine the interrelation between PLR and SSEP. PLR will be assessed by Neurological Pupil index (NPi) and SSEP by the cortical N20 response to stimulation of the median nerve.

DETAILED DESCRIPTION:
Background:

Anoxic/ischemic brain injury is the most common cause of death among comatose survivors of cardiac arrest (CA). The neurological prognosis of these patients is assessed using the multimodal prognostication model, which includes several methods. Somatosensory Evoked Potentials (SSEP) and Pupillary Light Reflex (PLR) are key methods for prognostication, as both have low false positive rates. Though they assess different functions of the brain, they should both be sensitive to severe anoxic/ischemic injury from cardiac arrest. The primary aim of the study is to describe the association between PLR quantified as the Neurological Pupil index (NPi) and bilateral absence of the cortical SSEP signal in patients remaining comatose after cardiac arrest. The secondary aim is to define a NPi cut-off value that renders a false positive rate (FPR) of less than 5% for a bilaterally absent SSEP response.

Methods:

An explorative, prospective, observational, cohort of 50 adult (>18 years) comatose survivors of CA admitted to the intensive care unit at Sahlgrenska University Hospital. The results from routine SSEP performed > 48 hours after CA and PLR assessed using NPi calculated by automated pupillometry are compared. Neurological outcome at hospital discharge is classified using the modified Rankin Scale (mRS), where poor neurological outcome is defined by mRS 4-6.

Statistical analysis:

In order to find a significant difference in NPi of 0.7 with a power of 95% with two-sided Fisher's non-parametric permutation test, 45 patients are needed assuming allocation 2:1 and unequal SD in the groups 0.37 and 0.67, calculated from the IQR above, and significance level 0.01. To account for uncertainty within these estimates, we aim to include 50 patients with a complete protocol.

A receiver operating characteristics curve (ROC-curve) will be used to find the NPi cut-off values resulting in a false positive rate of less than 5% for absent SSEP to predict poor neurological outcome. NPi values below the cut-off i.e., values consistent with poor outcome, will be used to calculate the predictive value for SSEP at its given prevalence. Fisher's exact test will be used to assess correlation between NPi and SSEP.

Discussion:

A clear correlation between the absence of cortical SSEP response and NPi values will permit application of the adequate method to the individual patient. This may also enable rationalisation of the multimodal assessment of the neurological prognosistication using a smaller number of methods. In clinical practice, this may render the prognostication of neurological function of comatose patients after cardiac arrest more accurate, as well as more cost- and time efficient.

ELIGIBILITY:
Inclusion Criteria:

>18-year-old comatose survivors of cardiac arrest with Glasgow coma scale < 9.

Exclusion Criteria:

return of consciousness before SSEP is performed; pregnancy; intracranial bleeding; traumatic brain injury; palliative care and lack of next of kin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 year old) comatose survivors of cardiac arrest admitted to the central intensive care unit at Sahlgrenska University Hospital in Gothenburg, Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The association between NPi and bilateral absence of the cortical SSEP response. | SSEP and pupillometry performed 48 hours after cardiac arrest
  ROC curve analysis

SECONDARY OUTCOMES:
NPi cut-off value that renders a false positive rate (FPR) of less than 5% for a bilaterally absent SSEP response. | SSEP and pupillometry performed 48 hours after cardiac arrest
  Analysed by stepwise crosstabulation of NPi values against absent cortical SSEP response.

OTHER OUTCOMES:
Predictive capacity for SSEP and NPi for death at 30 days and neurological outcome at hospital discharge | Assessed from medical records within a month after cardiac arrest
  Analysed as sensitivity, specificity and odds ratio

CONTACTS AND LOCATIONS:
Locations (1):
- avd 96 CIVA Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lilja L, Thuccani M, Joelsson S, Nilsson J, Redfors P, Lundgren P, Rylander C. The capacity of neurological pupil index to predict absence of somatosensory evoked potentials after cardiac arrest-A study protocol. Acta Anaesthesiol Scand. 2021 Jul;65(6):852-858. doi: 10.1111/aas.13822. Epub 2021 Mar 29. PMID 33735459